CLINICAL TRIAL: NCT01952678
Title: A Retrospective Clinical Study to Compare the Rates of Agreement Between Clinical Diagnosis and Visual Assessment of DaTscan™ Images in Non-Caucasian and Caucasian Subjects With Parkinson's Disease (PD) or Essential Tremor (ET)
Brief Title: Compare Rates of Agreement Between Clinical Diagnosis and Visual Assessment of DaTscan™ Images in Non-Caucasian and Caucasian Subjects With Parkinson's Disease (PD) or Essential Tremor (ET)
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: H2O Clinical LLC (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-001-011
Record Dates: First submitted 2013-09-19; First posted 2013-09-30 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2017-10

CONDITIONS: Essential Tremor; Parkinson's Disease
Keywords: DaTscan; Parkinson's Disease
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DaTscan™ - Non-Caucasian Participants: Non-Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
  Interventions: Other: DaTscan™ - Non-Caucasian Participants
- DaTscan™- Caucasian Participants: Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
  Interventions: Other: DaTscan™ - Caucasian Participants

INTERVENTIONS:
Other: DaTscan™ - Non-Caucasian Participants — Participants who previously administered DaTscan™ and had undergone SPECT imaging of the brain per local practice at each institution.
  Groups: DaTscan™ - Non-Caucasian Participants
Other: DaTscan™ - Caucasian Participants — Participants who previously administered DaTscan™ and had undergone SPECT imaging of the brain per local practice at each institution.
  Groups: DaTscan™- Caucasian Participants

SUMMARY:
The primary objective of this study is to determine if the diagnostic performance of DaTscan™ single photon emission computed tomography (SPECT) imaging is different in non-Caucasian subjects compared with Caucasian subjects with movement disorders.

ELIGIBILITY:
Inclusion Criteria:

For Non-Caucasians:

* Non-Caucasian male and female adult participants (greater than or equal to 18 years of age) with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
* The participant had existing diagnostic-quality and interpretable DaTscan SPECT images of the brain.

For Caucasians:

* Caucasian male and female adult participants (greater than or equal to 18 years of age) with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
* The participant had existing diagnostic-quality and interpretable DaTscan SPECT images of the brain.
* The participant was matched by final clinical diagnosis, sex and age (±5 years) with a non-Caucasian participant.

Exclusion Criteria:

* Known/suspected structural abnormalities of the brain (e.g., hydrocephalus; brain tumor; stroke; etc.) that could grossly distort the DaTscan images.
* Participants whose race and ethnic information could not be determined from source document review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-Caucasian and Caucasian Subjects With Parkinson's Disease (PD) or Essential Tremor (ET).
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2013-07-30; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Zubeldia, M.D., Study Chair — GE Healthcare
Locations (1):
- GE Healthcare, Marlborough, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the present study GE-001-011 (NCT01952678), participants who previously administered DaTscan™ and had undergone single photon emission computed tomography (SPECT) imaging of the brain per local practice at each institution, were enrolled.
Pre-assignment Details: A total of 102 non-Caucasian and 102 Caucasian participants were enrolled in the study.
Groups:
- DaTscan™- Non-Caucasian Participant: Non-Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected Parkinson's disease (PD) or Essential tremor (ET) who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
Period: Overall Study
Arm/Group | DaTscan™- Non-Caucasian Participant | DaTscan™- Caucasian Participants
Started | 102 | 102
Completed | 102 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants.
Groups:
- DaTscan™- Non-Caucasian Participants: Non-Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
- Total: Total of all reporting groups
Arm/Group | DaTscan™- Non-Caucasian Participants | DaTscan™- Caucasian Participants | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (11.09) | 66.4 (10.67) | 66.4 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 94
  Male | 55 | 55 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 94 | 93 | 187
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 28 | 0 | 28
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 66 | 0 | 66
  White | 0 | 102 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Positive Percent Agreement of Blinded Visual Assessment of Each Participant's DaTscan Image - Intent-to-diagnose (ITD) Population
Description: The majority blinded visual interpretation of each participant's image (3 blinded readers) was compared to his/her final clinical diagnosis, and the image interpretation was classified as true positive, false positive, true negative, or false negative. The counts of each classification type were used to determine the positive percent agreement (PPA, analogous to sensitivity) of the blinded visual image interpretations. The majority assessment was based on ≥ 2 of the 3 readers in agreement on the assessment.
Time Frame: Day 1
Population: ITD population that included all participants who underwent SPECT imaging after receiving DaTscan™ and enrolled in the study. Here, number of participants analyzed = participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Positive percent agreement
Groups:
- DaTscan™ - Non-Caucasian Participants: Non-Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging and had a final clinical diagnosis of PD.
- DaTscan™ - Caucasian Participants: Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging and had a final clinical diagnosis of PD.
Arm/Group | DaTscan™ - Non-Caucasian Participants | DaTscan™ - Caucasian Participants
Number analyzed (Participants) | 58 | 58
Positive percent agreement
  Reader A: number analyzed (Participants) | 57 | 57
  Reader A | 86.0 [74.2 to 93.7] | 84.2 [72.1 to 92.5]
  Reader B: number analyzed (Participants) | 57 | 57
  Reader B | 78.9 [66.1 to 88.6] | 86.0 [74.2 to 93.7]
  Reader C: number analyzed (Participants) | 57 | 57
  Reader C | 89.5 [78.5 to 96.0] | 87.7 [76.3 to 94.9]
  Majority: number analyzed (Participants) | 57 | 57
  Majority | 87.7 [76.3 to 94.9] | 86.0 [74.2 to 93.7]
Statistical Analysis 1: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader A: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.8, 95% CI 2-sided [-17.3 to 20.7]
Statistical Analysis 2: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader B: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 0.4608, Fisher Exact; Mean Difference (Net) = -7.0, 95% CI 2-sided [-25.8 to 12.1]
Statistical Analysis 3: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader C: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.8, 95% CI 2-sided [-17.3 to 20.7]
Statistical Analysis 4: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Majority Read: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.8, 95% CI 2-sided [-17.3 to 20.7]

2. Primary Outcome: Positive Percent Agreement of Blinded Visual Assessment of Each Participant's DaTscan Image - Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: Day 1
Population: PP population consisted of all participants who met inclusion/exclusion criteria, had DaTscan™ image sets that were considered evaluable by ≥2 of the 3 blinded readers, and had no major protocol violations from any of the matched pair participants. Here, number of participants analyzed = participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Positive percent agreement
Groups:
- DaTscan™ - Non-Caucasian Participants: Non-Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging, were included in PP population and had a final clinical diagnosis of PD.
- DaTscan™ - Caucasian Participants: Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging, were included in PP population and had a final clinical diagnosis of PD.
Arm/Group | DaTscan™ - Non-Caucasian Participants | DaTscan™ - Caucasian Participants
Number analyzed (Participants) | 56 | 56
Positive percent agreement
  Reader A | 85.7 [73.8 to 93.6] | 83.9 [71.7 to 92.4]
  Reader B | 78.6 [65.6 to 88.4] | 85.7 [73.8 to 93.6]
  Reader C | 89.3 [78.1 to 96.0] | 87.5 [75.9 to 94.8]
  Majority | 87.5 [75.9 to 94.8] | 85.7 [73.8 to 93.6]
Statistical Analysis 1: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader A: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.8, 95% CI 2-sided [-17.5 to 20.9]
Statistical Analysis 2: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader B: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 0.4599, Fisher Exact; Mean Difference (Net) = -7.1, 95% CI 2-sided [-26.1 to 12.2]
Statistical Analysis 3: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader C: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.8, 95% CI 2-sided [-17.5 to 20.9]
Statistical Analysis 4: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Majority Read: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: PPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.8, 95% CI 2-sided [-17.5 to 20.9]

3. Primary Outcome: Negative Percent Agreement of Blinded Visual Assessment of Each Participant's DaTscan Image - Intent-to-diagnose (ITD) Population
Description: The majority blinded visual interpretation of each participant's image (3 blinded readers) was compared to his/her final clinical diagnosis, and the image interpretation was classified as true positive, false positive, true negative, or false negative. The counts of each classification type were used to determine the negative percent agreement (NPA, analogous to specificity) of the blinded visual image interpretations. The majority assessment was based on ≥ 2 of the 3 readers in agreement on the assessment.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Negative percent agreement
Groups:
- DaTscan™- Non-Caucasian Participants: Non-Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging and had a final clinical diagnosis of ET.
- DaTscan™- Caucasian Participants: Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging and had a final clinical diagnosis of ET.
Arm/Group | DaTscan™- Non-Caucasian Participants | DaTscan™- Caucasian Participants
Number analyzed (Participants) | 44 | 43
Negative percent agreement
  Reader A: number analyzed (Participants) | 43 | 43
  Reader A | 93.0 [80.9 to 98.5] | 93.0 [80.9 to 98.5]
  Reader B | 84.1 [69.9 to 93.4] | 83.7 [69.3 to 93.2]
  Reader C | 86.4 [72.6 to 94.8] | 88.4 [74.9 to 96.1]
  Majority | 88.6 [75.4 to 96.2] | 88.4 [74.9 to 96.1]
Statistical Analysis 1: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader A: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 0.0, 95% CI 2-sided [-22.0 to 22.0]
Statistical Analysis 2: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader B: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 0.4, 95% CI 2-sided [-20.8 to 20.8]
Statistical Analysis 3: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader C: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = -2.0, 95% CI 2-sided [-23.0 to 18.5]
Statistical Analysis 4: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Majority Read: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 0.3, 95% CI 2-sided [-20.8 to 20.8]

4. Primary Outcome: Negative Percent Agreement of Blinded Visual Assessment of Each Participant's DaTscan Image - Per Protocol (PP) Population
Description: as for outcome 3
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Negative percent agreement
Groups:
- DaTscan™ - Non-Caucasian Participants: Non-Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging, were included in PP population and had a final clinical diagnosis of ET.
- DaTscan™ - Caucasian Participants: Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging, were included in PP population and had a final clinical diagnosis of ET.
Arm/Group | DaTscan™ - Non-Caucasian Participants | DaTscan™ - Caucasian Participants
Number analyzed (Participants) | 41 | 40
Negative percent agreement
  Reader A: number analyzed (Participants) | 40 | 40
  Reader A | 92.5 [79.6 to 98.4] | 92.5 [79.6 to 98.4]
  Reader B | 90.2 [76.9 to 97.3] | 85.0 [70.2 to 94.3]
  Reader C | 90.2 [76.9 to 97.3] | 90.0 [76.3 to 97.2]
  Majority | 92.7 [80.1 to 98.5] | 90.0 [76.3 to 97.2]
Statistical Analysis 1: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader A: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 0.0, 95% CI 2-sided [-22.8 to 22.8]
Statistical Analysis 2: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader B: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 0.5187, Fisher Exact; Mean Difference (Net) = 5.2, 95% CI 2-sided [-16.7 to 26.2]
Statistical Analysis 3: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Reader C: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 0.2, 95% CI 2-sided [-21.5 to 21.5]
Statistical Analysis 4: Comparison: DaTscan™ - Non-Caucasian Participants vs DaTscan™ - Caucasian Participants; Majority Read: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: NPA was equal for Caucasian and non-Caucasian populations; p = 0.7123, Fisher Exact; Mean Difference (Net) = 2.7, 95% CI 2-sided [-19.1 to 23.9]

5. Secondary Outcome: Overall Percent Agreement of Blinded Visual Assessment of Each Participant's DaTscan Image - Intent-to-diagnose (ITD) Population
Description: Overall percent agreement (OPA) regardless of image interpretation (analogous to accuracy; ratio of number of true results / number of all participants) for each racial group, was tested to determine if it was greater than 80% in both racial groups. The majority assessment was based on ≥2 of the 3 readers in agreement on the assessment.
Time Frame: Day 1
Population: The intent-to-diagnose (ITD) population that included all participants who underwent SPECT imaging after receiving DaTscan™ and enrolled in the study. Here, number of participants analyzed = participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Overall percent agreement
Arm/Group | DaTscan™- Non-Caucasian Participants | DaTscan™- Caucasian Participants
Number analyzed (Participants) | 101 | 100
Overall percent agreement
  Reader A: number analyzed (Participants) | 100 | 100
  Reader A | 89.0 [81.2 to 94.4] | 88.0 [80.0 to 93.6]
  Reader B | 81.2 [72.2 to 88.3] | 85.0 [76.5 to 91.4]
  Reader C | 88.1 [80.2 to 93.7] | 88.0 [80.0 to 93.6]
  Majority | 88.1 [80.2 to 93.7] | 87.0 [78.8 to 92.9]
Statistical Analysis 1: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader A: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.0, 95% CI 2-sided [-13.3 to 15.3]
Statistical Analysis 2: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader B: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 0.5731, Fisher Exact; Mean Difference (Net) = -3.8, 95% CI 2-sided [-17.7 to 9.8]
Statistical Analysis 3: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader C: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 0.1, 95% CI 2-sided [-13.8 to 13.8]
Statistical Analysis 4: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Majority Read: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 0.8340, Fisher Exact; Mean Difference (Net) = 1.1, 95% CI 2-sided [-12.8 to 14.7]

6. Secondary Outcome: Overall Percent Agreement of Blinded Visual Assessment of Each Participant's DaTscan Image - Per Protocol (PP) Population
Description: as for outcome 5
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Overall percent agreement
Groups:
- DaTscan™- Non-Caucasian Participants: Non-Caucasian participants previously administered DaTscan™, included in PP population with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
- DaTscan™- Caucasian Participants: Caucasian participants previously administered DaTscan™, included in PP population with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
Arm/Group | DaTscan™- Non-Caucasian Participants | DaTscan™- Caucasian Participants
Number analyzed (Participants) | 97 | 96
Overall percent agreement
  Reader A: number analyzed (Participants) | 96 | 96
  Reader A | 88.5 [80.4 to 94.1] | 87.5 [79.2 to 93.4]
  Reader B | 83.5 [74.6 to 90.3] | 85.4 [76.7 to 91.8]
  Reader C | 89.7 [81.9 to 94.9] | 88.5 [80.4 to 94.1]
  Majority | 89.7 [81.9 to 94.9] | 87.5 [79.2 to 93.4]
Statistical Analysis 1: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader A: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 1.0000, Fisher Exact; Mean Difference (Net) = 1.0, 95% CI 2-sided [-13.5 to 15.6]
Statistical Analysis 2: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader B: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 0.8429, Fisher Exact; Mean Difference (Net) = -1.9, 95% CI 2-sided [-16.1 to 12.0]
Statistical Analysis 3: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Reader C: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 0.8214, Fisher Exact; Mean Difference (Net) = 1.1, 95% CI 2-sided [-13.0 to 15.0]
Statistical Analysis 4: Comparison: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Majority Read: DaTscan™- Non-Caucasian Participants vs DaTscan™- Caucasian Participants; Test type: Equivalence — Analysis was performed using the hypothesis: OPA was equal for Caucasian and non-Caucasian populations; p = 0.6577, Fisher Exact; Mean Difference (Net) = 2.2, 95% CI 2-sided [-12.0 to 16.1]

ADVERSE EVENTS:
Description: As the present study GE-001-011 was a retrospective study, therefore, no safety evaluations performed in this study.
Groups:
- DaTscan™ - Caucasian Participants: Caucasian participants previously administered DaTscan™, with an initial diagnosis of suspected PD or ET who underwent DaTscan SPECT imaging to assist with the participant's final clinical diagnosis of PD or ET.
Arm/Group | DaTscan™- Non-Caucasian Participants | DaTscan™ - Caucasian Participants
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.